CLINICAL TRIAL: NCT02608177
Title: Continuous Glucose Monitoring to Assess Glycemia in Chronic Kidney Disease - Changing Glucose Management
Acronym: CANDY-CANE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: American Diabetes Association (Other); Medtronic (Industry); Abbott (Industry)
Responsible Party: Principal Investigator, Ian deBoer, Associate Professor, Medicine/Nephrology, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 50084
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Results first posted 2018-09-13 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-08

CONDITIONS: Chronic Kidney Diseases; Type 2 Diabetes
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — Linagliptin; Glipizide

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Linagliptin/Glipizide (Experimental): Arm receives 4 weeks of study drug linagliptin followed by 4 weeks of glipizide
  Interventions: Drug: Linagliptin; Drug: Glipizide
- Glipizide/Linagliptin (Experimental): Arm receives 4 weeks of study drug glipizide followed by 4 weeks linagliptin
  Interventions: Drug: Linagliptin; Drug: Glipizide

INTERVENTIONS:
Drug: Linagliptin — Receives 4 weeks of study drug linagliptin
Drug: Glipizide — Receives 4 weeks of study drug glipizide

SUMMARY:
The goal of this study is to test whether a dipeptidyl peptidase-4 inhibitor, compared with a sulfonylurea, improves time in normal blood glucose range and reduces blood glucose variability. Blood glucose is measured using a continuous glucose monitoring device.

DETAILED DESCRIPTION:
This is a proof-of-concept clinical trial testing the effects of linagliptin versus glipizide on glucose variability among people with type 2 diabetes and stage 3-4 CKD. In a cross-over design, each enrolled participant will receive 28 days of each study medication. Study medications will be provided in a randomly assigned order without blinding. The primary study outcome is glucose time in range, measured by blinded continuous glucose monitoring for the last 6 days of each 28-day treatment period. Secondary outcomes include indices of glycemic variability, hypoglycemia, and biomarkers of systemic inflammation, oxidative stress, and albuminuria. The overall goal of this research is to identify safe and effective treatments to control glycemia among patients with diabetes and CKD.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* eGFR 15-59 mL/min/1.73 m2
* Hemoglobin A1c < 8%
* Age ≥ 18 years
* Current use of sulfonylurea

Exclusion Criteria:

* BMI > 40 kg/m2
* Actively using CGM for clinical care
* End stage renal disease needing dialysis
* Kidney transplant
* Pregnant or nursing
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-11; Primary Completion 2017-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian de Boer, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Linagliptin/Glipizide | Glipizide/Linagliptin
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Linagliptin/Glipizide | Glipizide/Linagliptin | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (9.9) | 70.4 (NA) — no SD due to one participant enrolled | 68.3 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic white race/ethnicity | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Glucose Time in Range
Description: Time with glucose 70-140 mg/dL
Time Frame: last 6 days of each 28-day treatment period
Measure: Mean (Standard Deviation); unit: minutes per day
Groups:
- Glipizide: Outcome assessed among all participants in both treatment groups at the end of treatment with Glipizide for 4 weeks.
- Linagliptin: Outcome assessed among all participants in both treatment groups at the end of treatment with Linagliptin for 4 weeks.
Arm/Group | Glipizide | Linagliptin
Number analyzed (Participants) | 3 | 3
minutes per day | 495.2 (671.9) | 573.3 (669.1)

2. Secondary Outcome: Glycemic Variability
Description: SD of glucose readings
Time Frame: last 6 days of each 28-day treatment period
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Glipizide | Linagliptin
Number analyzed (Participants) | 3 | 3
mg/dL | 40.9 (16.1) | 41.5 (22.7)

3. Secondary Outcome: Hypoglycemia
Description: Glucose <70 mg/dL for at least 10 minutes
Time Frame: last 6 days of each 28-day treatment period
Measure: Number; unit: events
Arm/Group | Glipizide | Linagliptin
Number analyzed (Participants) | 3 | 3
events | 4 | 2

4. Secondary Outcome: Biomarkers of Systemic Inflammation
Description: Measured by plasma C-reactive protein (CRP)
Time Frame: last 6 days of each 28-day treatment period
Population: Labs not run due to small sample size.
Arm/Group | Linagliptin/Glipizide | Glipizide/Linagliptin
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Biomarkers of Systemic Inflammation
Description: Measured by plasma interleukin-6
Time Frame: last 6 days of each 28-day treatment period
Population: Labs not run due to small sample size.
Arm/Group | Linagliptin/Glipizide | Glipizide/Linagliptin
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Biomarkers of Oxidative Stress
Description: Measured by plasma F2-isoprostanes
Time Frame: last 6 days of each 28-day treatment period
Population: Labs not run due to small sample size.
Arm/Group | Linagliptin/Glipizide | Glipizide/Linagliptin
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Biomarkers of Oxidative Stress
Description: Measured by urine F2-isoprostanes
Time Frame: last 6 days of each 28-day treatment period
Population: Labs not run due to small sample size.
Arm/Group | Linagliptin/Glipizide | Glipizide/Linagliptin
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Biomarkers of Albuminuria
Description: Measured by albumin-creatinine ratio
Time Frame: last 6 days of each 28-day treatment period
Population: Labs not run due to small sample size.
Arm/Group | Linagliptin/Glipizide | Glipizide/Linagliptin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: AE information collected over 8 weeks of the study
Arm/Group | Linagliptin/Glipizide | Glipizide/Linagliptin
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT02608177/Prot_SAP_000.pdf